CLINICAL TRIAL: NCT00278694
Title: Oxaliplatin and 5-FU Based Preoperative Chemoradiation
Acronym: LARC-RRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, Senior consultant medical oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-05059; Eudractnr 2005-000024-16
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Cancer
Keywords: Oxaliplatin, radiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Chemoradiotherapy; Fluorouracil

ARMS (1):
- Chemoradiation (Experimental): Neoadjuvant chemotherapy and chemoradiation
  Interventions: Drug: Oxaliplatin; Drug: Chemoradiation; Drug: 5-FU; Radiation: Preoperative chemoradiation; Procedure: Pelvic surgery; Drug: Neoadjuvant oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin
Drug: Chemoradiation
Drug: 5-FU
Radiation: Preoperative chemoradiation
Procedure: Pelvic surgery
Drug: Neoadjuvant oxaliplatin

SUMMARY:
Oxaliplatin and 5FU based preoperative chemoradiation in rectal cancer.

DETAILED DESCRIPTION:
Effect of treatment, safety profile and quality of life scorings.

ELIGIBILITY:
Rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2005-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety profile | 5 years
Number of patients obtaining pCR | 5 years

SECONDARY OUTCOMES:
Clinical, radiological and molecular response to treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Georg Høyer, DH, Study Chair — South region committee for research ethics in Norway
Locations (1):
- RRHF, Oslo, Norway

REFERENCES:
- [Derived] Abrahamsson H, Porojnicu AC, Lindstrom JC, Dueland S, Flatmark K, Hole KH, Seierstad T, Moan J, Redalen KR, Meltzer S, Ree AH. High level of circulating vitamin D during neoadjuvant therapy may lower risk of metastatic progression in high-risk rectal cancer. BMC Cancer. 2019 May 23;19(1):488. doi: 10.1186/s12885-019-5724-z. PMID 31122213
- [Derived] Kalanxhi E, Hektoen HH, Meltzer S, Dueland S, Flatmark K, Ree AH. Circulating proteins in response to combined-modality therapy in rectal cancer identified by antibody array screening. BMC Cancer. 2016 Jul 26;16:536. doi: 10.1186/s12885-016-2601-x. PMID 27461255
- [Derived] Hektoen HH, Flatmark K, Andersson Y, Dueland S, Redalen KR, Ree AH. Early increase in circulating carbonic anhydrase IX during neoadjuvant treatment predicts favourable outcome in locally advanced rectal cancer. BMC Cancer. 2015 Jul 24;15:543. doi: 10.1186/s12885-015-1557-6. PMID 26205955
- [Derived] Ree AH, Flatmark K, Saelen MG, Folkvord S, Dueland S, Geisler J, Redalen KR. Tumor phosphatidylinositol 3-kinase signaling in therapy resistance and metastatic dissemination of rectal cancer: opportunities for signaling-adapted therapies. Crit Rev Oncol Hematol. 2015 Jul;95(1):114-24. doi: 10.1016/j.critrevonc.2015.01.003. Epub 2015 Jan 12. PMID 25624177